CLINICAL TRIAL: NCT06855498
Title: A Phase 3b, Multicenter, Rollover Study for Participants Previously Enrolled in Clinical Trials of Povorcitinib
Brief Title: Rollover Study for Participants Previously Enrolled in Clinical Trials of Povorcitinib
Acronym: STOP-LTR
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INCB054707-801; 2024-520107-12-00 (Registry Identifier: EU CT Number)
Record Dates: First submitted 2025-02-26; First posted 2025-03-03 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Hidradenitis Suppurativa (HS)
Keywords: INCB054707; povorcitinib; Hidradenitis Suppurativa; Hidradenitis; HS
MeSH Terms: conditions — Hidradenitis Suppurativa; Hidradenitis

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- povorcitinib (Experimental): Participants will receive povorcitinib treatment with the same schedule and dose options as the study in which they originally enrolled.
  Interventions: Drug: povorcitinib

INTERVENTIONS:
Drug: povorcitinib — Study drug will be taken orally as defined by the protocol.

SUMMARY:
Rollover study for participants from predetermined, Incyte-sponsored parent clinical trials of povorcitinib.

ELIGIBILITY:
Inclusion Criteria:

* Ability to comprehend and willingness to sign a written ICF for the study.
* Completed the treatment period of a predetermined, Incyte-sponsored, povorcitinib parent study without safety or tolerability concerns, per investigator's assessment.
* Received clinical benefit from treatment with study drug during the parent study, as determined by the investigator.
* Demonstrated compliance, as assessed by the investigator, with the parent Protocol requirements.
* Willingness to avoid pregnancy or fathering children as defined in the protocol.
* Willingness and ability to comply with the study Protocol and procedures.

Exclusion Criteria:

* Had been permanently discontinued from study treatment during the parent study.
* Had temporary study drug interruption due to safety and/or efficacy reasons at or after the final visit of the parent study.
* Received at least 1 dose of either of the following therapies within the 28 days prior to starting treatment in this rollover study:

  * Biologic immunomodulator (examples include but are not limited to adalimumab, bimekizumab, dupilumab, infliximab, nemolizumab, secukinumab).
  * Live, attenuated vaccine.
* Plans for administration of a live, attenuated vaccine during this study or within 8 weeks after the last dose of study drug.
* Women who are pregnant (or who are considering pregnancy) or breastfeeding.
* Known hypersensitivity or severe reaction to povorcitinib or excipients of povorcitinib and/or other products in the same class.
* Currently enrolled in any other clinical study involving an investigational product or any other type of medical research judged not to be scientifically or medically compatible with this study.
* Any condition that would, in the investigator's and/or sponsor's judgment, interfere with full participation in the study, including administration of study drug and attending required study visits; pose a significant risk to the participant; or interfere with interpretation of study data.

Other protocol-defined Inclusion/Exclusion Criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2025-02-28 (Actual); Primary Completion 2028-02-28 (Estimated); Study Completion 2028-02-28 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants with Treatment-Emergent Adverse Events (TEAEs) | Up to approximately 3 years
  Adverse events either reported for the first time in this Protocol or any AE ongoing and defined as treatment-emergent from the parent Protocol.

SECONDARY OUTCOMES:
Proportion of participants with a total ANdT count of 0, 1, or 2 at each visit | Up to approximately 3 years
  ANdT count is defined as the total sum of abscesses, inflammatory nodules, and draining tunnels.

CONTACTS AND LOCATIONS:
Overall Officials: Incyte Medical Monitor, Study Director — Incyte Corporation
Locations (329):
- United States (111):
  - Investigative Site US086, Birmingham, Alabama
  - Investigative Site US098, Montgomery, Alabama
  - Investigative Site US004, Phoenix, Arizona
  - Investigative Site US047, Scottsdale, Arizona
  - Investigative Site US124, Scottsdale, Arizona
  - Investigative Site US115, Tucson, Arizona
  - Investigative Site US113, Fayetteville, Arkansas
  - Investigative Site US045, Fort Smith, Arkansas
  - Investigative Site US110, Hot Springs, Arkansas
  - Investigative Site US009, Rogers, Arkansas
  - Investigative Site US076, Fountain Valley, California
  - Investigative Site US077, Fremont, California
  - Investigative Site US071, Huntington Beach, California
  - Investigative Site US020, Laguna Niguel, California
  - Investigative Site US036, Los Angeles, California
  - Investigative Site US067, Los Angeles, California
  - Investigative Site US060, Northridge, California
  - Investigative Site US037, Oakland, California
  - Investigative Site US089, Santa Monica, California
  - Investigative Site US080, Sherman Oaks, California
  - Investigative Site US129, Aventura, Florida
  - Investigative Site US116, Boca Raton, Florida
  - Investigative Site US002, Boca Raton, Florida
  - Investigative Site US062, Coral Gables, Florida
  - Investigative Site US084, Coral Gables, Florida
  - Investigative Site US017, Hialeah, Florida
  - Investigative Site US019, Hollywood, Florida
  - Investigative Site US090, Hollywood, Florida
  - Investigative Site US044, Margate, Florida
  - Investigative Site US015, Miami, Florida
  - Investigative Site US059, Miami, Florida
  - Investigative Site US072, Miami Lakes, Florida
  - Investigative Site US079, Miami Lakes, Florida
  - Investigative Site US023, North Miami Beach, Florida
  - Investigative Site US029, Ocala, Florida
  - Investigative Site US133, Tampa, Florida
  - Investigative Site US035, Tampa, Florida
  - Investigative Site US005, Tampa, Florida
  - Investigative Site US001, Tampa, Florida
  - Investigative Site US066, West Palm Beach, Florida
  - Investigative Site US070, West Palm Beach, Florida
  - Investigative Site US051, Marietta, Georgia
  - Investigative Site US103, Sandy Springs, Georgia
  - Investigative Site US100, Stonecrest, Georgia
  - Investigative Site US125, Chicago, Illinois
  - Investigative Site US093, Chicago, Illinois
  - Investigative Site US049, Skokie, Illinois
  - Investigative Site US039, West Dundee, Illinois
  - Investigative Site US112, Clarksville, Indiana
  - Investigative Site US108, Indianapolis, Indiana
  - Investigative Site US008, Indianapolis, Indiana
  - Investigative Site US064, West Lafayette, Indiana
  - Investigative Site US056, Bowling Green, Kentucky
  - Investigative Site US012, Baton Rouge, Louisiana
  - Investigative Site US057, New Orleans, Louisiana
  - Investigative Site US111, Baltimore, Maryland
  - Investigative Site US038, Baltimore, Maryland
  - Investigative Site US099, Glenn Dale, Maryland
  - Investigative Site US053, Marriottsville, Maryland
  - Investigative Site US101, Rockville, Maryland
  - Investigative Site US127, Rockville, Maryland
  - Investigative Site US030, Boston, Massachusetts
  - Investigative Site US048, Brighton, Massachusetts
  - Investigative Site US061, Ann Arbor, Michigan
  - Investigative Site US114, Auburn Hills, Michigan
  - Investigative Site US120, Detroit, Michigan
  - Investigative Site US091, Troy, Michigan
  - Investigative Site US128, Troy, Michigan
  - Investigative Site US042, Waterford, Michigan
  - Investigative Site US011, Minneapolis, Minnesota
  - Investigative Site US088, Saint Joseph, Missouri
  - Investigative Site US016, St Louis, Missouri
  - Investigative Site US096, Las Vegas, Nevada
  - Investigative Site US007, Portsmouth, New Hampshire
  - Investigative Site US121, Hackensack, New Jersey
  - Investigative Site US118, Albuquerque, New Mexico
  - Investigative Site US082, East Syracuse, New York
  - Investigative Site US123, East Syracuse, New York
  - Investigative Site US040, Kew Gardens, New York
  - Investigative Site US034, New York, New York
  - Investigative Site US081, New York, New York
  - Investigative Site US065, New York, New York
  - Investigative Site US075, New York, New York
  - Investigative Site US050, Rochester, New York
  - Investigative Site US131, Stony Brook, New York
  - Investigative Site US031, Chapel Hill, North Carolina
  - Investigative Site US028, Bexley, Ohio
  - Investigative Site US055, Boardman, Ohio
  - Investigative Site US025, Cincinnati, Ohio
  - Investigative Site US073, Columbus, Ohio
  - Investigative Site US033, Columbus, Ohio
  - Investigative Site US130, Dayton, Ohio
  - Investigative Site US117, Dublin, Ohio
  - Investigative Site US085, Oklahoma City, Oklahoma
  - Investigative Site US074, Philadelphia, Pennsylvania
  - Investigative Site US069, Plymouth Meeting, Pennsylvania
  - Investigative Site US119, Yardley, Pennsylvania
  - Investigative Site US021, Bellaire, Texas
  - Investigative Site US078, Dallas, Texas
  - Investigative Site US010, Dallas, Texas
  - Investigative Site US054, Pflugerville, Texas
  - Investigative Site US083, San Antonio, Texas
  - Investigative Site US126, Sugar Land, Texas
  - Investigative Site US068, Webster, Texas
  - Investigative Site US122, Murray, Utah
  - Investigative Site US063, South Jordan, Utah
  - Investigative Site US027, Norfolk, Virginia
  - Investigative Site US094, Richmond, Virginia
  - Investigative Site US132, Mill Creek, Washington
  - Investigative Site US092, Seattle, Washington
  - Investigative Site US003, Spokane, Washington
- Argentina (6):
  - Investigative Site AR005, Buenos Aires
  - Investigative Site AR002, Buenos Aires
  - Investigative Site AR006, Buenos Aires
  - Investigative Site AR004, Mar del Plata
  - Investigative Site AR003, Rosario
  - Investigative Site AR001, San Miguel de Tucumán
- Australia (11):
  - Investigative Site AU001, Charleston, New South Wales
  - Investigative Site AU003, Kogarah, New South Wales
  - Investigative Site AU005, Liverpool, New South Wales
  - Investigative Site AU010, Sydney, New South Wales
  - Investigative Site AU007, Wolloongabba, Queensland
  - Investigative Site AU006, Woolloongabba, Queensland
  - Investigative Site AU004, Carlton, Victoria
  - Investigative Site AU002, Melbourne, Victoria
  - Investigative Site AU011, Melbourne, Victoria
  - Investigative Site AU008, Fremantle
  - Investigative Site AU009, Westmead
- Austria (3):
  - Investigative Site AT002, Graz
  - Investigative Site AT004, Innsbruck
  - Investigative Site AT003, Vienna
- Belgium (6):
  - Investigative Site BE007, Bruges
  - Investigative Site BE002, Brussels
  - Investigative Site BE001, Ghent
  - Investigative Site BE003, Liège
  - Investigative Site BE006, Loverval
  - Investigative Site BE005, Woluwe-Saint-Lambert
- Bulgaria (14):
  - Investigative Site BG008, Dupnitsa
  - Investigative Site BG010, Lovech
  - Investigative Site BG012, Pleven
  - Investigative Site BG013, Plovdiv
  - Investigative Site BG007, Sevlievo
  - Investigative Site BG009, Sofia
  - Investigative Site BG002, Sofia
  - Investigative Site BG006, Sofia
  - Investigative Site BG011, Sofia
  - Investigative Site BG003, Sofia
  - Investigative Site BG001, Sofia
  - Investigative Site BG014, Sofia
  - Investigative Site BG005, Sofia
  - Investigative Site BG004, Stara Zagora
- Canada (28):
  - Investigative Site CA023, Calgary, Alberta
  - Investigative Site CA008, Calgary, Alberta
  - Investigative Site CA005, Edmonton, Alberta
  - Investigative Site CA028, Edmonton, Alberta
  - Investigative Site CA027, Edmonton, Alberta
  - Investigative Site CA013, Surrey, British Columbia
  - Investigative Site CA024, Vancouver, British Columbia
  - Investigative Site CA003, Winnipeg, Manitoba
  - Investigative Site CA006, Fredericton, New Brunswick
  - Investigative Site CA004, Barrie, Ontario
  - Investigative Site CA030, Cobourg, Ontario
  - Investigative Site CA011, Hamilton, Ontario
  - Investigative Site CA025, London, Ontario
  - Investigative Site CA002, London, Ontario
  - Investigative Site CA022, Markham, Ontario
  - Investigative Site CA014, Mississauga, Ontario
  - Investigative Site CA016, Mississauga, Ontario
  - Investigative Site CA001, Peterborough, Ontario
  - Investigative Site CA010, Richmond Hill, Ontario
  - Investigative Site CA017, Toronto, Ontario
  - Investigative Site CA018, Toronto, Ontario
  - Investigative Site CA021, Toronto, Ontario
  - Investigative Site CA019, Waterloo, Ontario
  - Investigative Site CA020, Québec, Quebec
  - Investigative Site CA026, Québec, Quebec
  - Investigative Site CA009, Saint-Jérôme, Quebec
  - Investigative Site CA029, Verdun, Quebec
  - Investigative Site CA015, Saskatoon, Saskatchewan
- Chile (3):
  - Investigative Site CL002, LAS Condes Santiago
  - Investigative Site CL003, Santiago
  - Investigative Site CL001, Valdivia
- Czechia (4):
  - Investigative Site CZ002, Ostrava-poruba
  - Investigative Site CZ004, Prague
  - Investigative Site CZ003, Prague
  - Investigative Site CZ001, Prague
- Denmark (2):
  - Investigative Site DK001, Aarhus
  - Investigative Site DK002, Roskilde
- France (15):
  - Investigative Site FR014, Antony
  - Investigative Site FR006, Bordeaux
  - Investigative Site FR004, Brest
  - Investigative Site FR015, Créteil
  - Investigative Site FR009, Lyon
  - Investigative Site FR012, Marseille
  - Investigative Site FR016, Mulhouse
  - Investigative Site FR011, Nantes
  - Investigative Site FR008, Nice
  - Investigative Site FR010, Paris
  - Investigative Site FR005, Reims
  - Investigative Site FR018, Romans-sur-Isère
  - Investigative Site FR007, Rouen
  - Investigative Site FR003, Saint-Priest-en-Jarez
  - Investigative Site FR001, Toulouse
- Germany (34):
  - Investigative Site DE036, Aachen
  - Investigative Site DE025, Bad Bentheim
  - Investigative Site DE005, Berlin
  - Investigative Site DE026, Berlin
  - Investigative Site DE006, Bochum
  - Investigative Site DE037, Bonn
  - Investigative Site DE024, Buxtehude
  - Investigative Site DE023, Chemnitz
  - Investigative Site DE013, Darmstadt
  - Investigative Site DE019, Darmstadt
  - Investigative Site DE027, Dortmund
  - Investigative Site DE012, Dresden
  - Investigative Site DE014, Düsseldorf
  - Investigative Site DE009, Erlangen
  - Investigative Site DE011, Frankfurt am Main
  - Investigative Site DE021, Friedrichshafen
  - Investigative Site DE010, Göttingen
  - Investigative Site DE032, Halle
  - Investigative Site DE001, Hamburg
  - Investigative Site DE002, Hanover
  - Investigative Site DE017, Heidelberg
  - Investigative Site DE003, Kiel
  - Investigative Site DE033, Leipzig
  - Investigative Site DE034, Lübeck
  - Investigative Site DE029, Magdeburg
  - Investigative Site DE022, Mahlow
  - Investigative Site DE015, Mainz
  - Investigative Site DE035, Mainz
  - Investigative Site DE038, Marburg
  - Investigative Site DE008, Merzig
  - Investigative Site DE030, München
  - Investigative Site DE028, Oldenburg
  - Investigative Site DE031, Tübingen
  - Investigative Site DE018, Witten
- Greece (3):
  - Investigative Site GR001, Athens
  - Investigative Site GR002, Athens
  - Investigative Site GR003, Thessaloniki
- Hungary (2):
  - Investigative Site HU001, Debrecen
  - Investigative Site HU002, Szombathely
- Italy (13):
  - Investigative Site IT012, Bari
  - Investigative Site IT009, Brescia
  - Investigative Site IT001, Catania
  - Investigative Site IT007, Chieti
  - Investigative Site IT014, Florence
  - Investigative Site IT010, L’Aquila
  - Investigative Site IT005, Milan
  - Investigative Site IT008, Naples
  - Investigative Site IT013, Perugia
  - Investigative Site IT006, Pisa
  - Investigative Site IT002, Rome
  - Investigative Site IT003, Rozzano
  - Investigative Site IT004, Torrette DI Ancona
- Netherlands (6):
  - Investigative Site NL005, Amsterdam
  - Investigative Site NL007, Amsterdam
  - Investigative Site NL006, Bergen op Zoom
  - Investigative Site NL003, Groningen
  - Investigative Site NL001, Rotterdam
  - Investigative Site NL004, Veldhoven
- Poland (29):
  - Investigative Site PL013, Cracov
  - Investigative Site PL009, Gdansk
  - Investigative Site PL029, Grodzisk Mazowiecki
  - Investigative Site PL011, Katowice
  - Investigative Site PL035, Kielce
  - Investigative Site PL031, Lublin
  - Investigative Site PL002, Lublin
  - Investigative Site PL020, Osielsko
  - Investigative Site PL006, Ostrowiec Świętokrzyski
  - Investigative Site PL016, Poznan
  - Investigative Site PL003, Rzeszów
  - Investigative Site PL015, Szczecin
  - Investigative Site PL028, Szczecin
  - Investigative Site PL041, Szczecin
  - Investigative Site PL010, Tarnów
  - Investigative Site PL030, Torun
  - Investigative Site PL017, Warsaw
  - Investigative Site PL026, Warsaw
  - Investigative Site PL007, Warsaw
  - Investigative Site PL014, Warsaw
  - Investigative Site PL012, Warsaw
  - Investigative Site PL004, Warsaw
  - Investigative Site PL027, Warsaw
  - Investigative Site PL024, Wrocaw
  - Investigative Site PL018, Wroclaw
  - Investigative Site PL001, Wroclaw
  - Investigative Site PL005, Wroclaw
  - Investigative Site PL008, Wroclaw
  - Investigative Site PL022, Wroclaw
- South Korea (8):
  - Investigative Site KR006, Ansan-si
  - Investigative Site KR008, Bucheon-si
  - Investigative Site KR007, Busan
  - Investigative Site KR003, Incheon
  - Investigative Site KR004, Jeonju
  - Investigative Site KR002, Seoul
  - Investigative Site KR005, Seoul
  - Investigative Site KR001, Yangsan
- Spain (16):
  - Investigative Site ES001, Badalona
  - Investigative Site ES010, Barcelona
  - Investigative Site ES017, Barcelona
  - Investigative Site ES015, Córdoba
  - Investigative Site ES003, Granada
  - Investigative Site ES013, Granada
  - Investigative Site ES006, Las Palmas de Gran Canaria
  - Investigative Site ES014, Madrid
  - Investigative Site ES008, Madrid
  - Investigative Site ES011, Madrid
  - Investigative Site ES012, Madrid
  - Investigative Site ES004, Manises
  - Investigative Site ES022, Pamplona
  - Investigative Site ES002, Santiago de Compostela
  - Investigative Site ES023, Santiago de Compostela
  - Investigative Site ES018, Valencia
- Switzerland (3):
  - Investigative Site CH003, Bern
  - Investigative Site CH001, Buochs
  - Investigative Site CH002, Zurich
- United Kingdom (12):
  - Investigative Site GB003, Birmingham
  - Investigative Site GB001, Dudley
  - Investigative Site GB011, Ipswich
  - Investigative Site GB002, Leeds
  - Investigative Site GB009, Leicester
  - Investigative Site GB013, Liverpool
  - Investigative Site GB012, London
  - Investigative Site GB014, London
  - Investigative Site GB006, Poole
  - Investigative Site GB007, Redhill
  - Investigative Site GB004, Salford
  - Investigative Site GB008, Wolverhampton

IPD SHARING:
Plan to Share IPD: Yes
Incyte shares data with qualified external researchers after a research proposal is submitted. These requests are reviewed and approved by a review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  The trial data availability is according to the criteria and process described on https://www.incyte.com/our-company/compliance-and-transparency
Supporting Information: Study Protocol, SAP
Time Frame: Data will be shared after the primary publication or 2 years after the study has ended for market authorized products and indications.
Access Criteria: Data from eligible studies will be shared with qualified researchers according to the criteria and process described in the Data Sharing section of the www.incyteclinicaltrials.com website. For approved requests, the researchers will be granted access to anonymized data under the terms of a data sharing agreement.
URL: https://www.incyte.com/our-company/compliance-and-transparency

REFERENCES:
- See also: Rollover Study for Participants Previously Enrolled in Clinical Trials of Povorcitinib — https://incyteclinicaltrials.com/studies/incb054707-801